CLINICAL TRIAL: NCT03638869
Title: A Phase 1 Study to Investigate the Safety, Tolerability, and Pharmacokinetic Profile of Multiple Ascending Doses of REL-1017 (d-Methadone) in Healthy Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of Multiple Ascending Doses of REL-1017 (d-Methadone)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Relmada Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: REL-1017-112
Record Dates: First submitted 2018-08-10; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — D-methadone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Placebo Comparator): 100 mL Ocean Spray® Diet Cranberry Juice
  Interventions: Drug: Placebo
- Arm 2 (Experimental): REL-1017 25 mg in 100 mL of Ocean Spray® Diet Cranberry Juice
  Interventions: Drug: REL-1017
- Arm 3 (Experimental): REL-1017 50 mg in 100 mL of Ocean Spray® Diet Cranberry Juice
  Interventions: Drug: REL-1017
- Arm 4 (Experimental): REL-1017 75 mg in 100 mL of Ocean Spray® Diet Cranberry Juice
  Interventions: Drug: REL-1017

INTERVENTIONS:
Drug: REL-1017 — The investigational product, REL-1017 is prepared as a solution with Ocean Spray® Diet Cranberry Juice on site to obtain a final volume of 100 mL for dosing. The study drug will be administered as a solution of 25 mg, 50 or 75 mg REL-1017 for 10 days, based on randomization prepared in Ocean Spray® Diet Cranberry Juice with a final volume of 100 mL.
  Other Names: (d-Methadone)
  Arms: Arm 2; Arm 3; Arm 4
Drug: Placebo
  Arms: Arm 1

SUMMARY:
This study evaluated the safety, tolerance, and pharmacokinetics (PK) of d-methadone in a limited dose range, in multiple administrations in humans.

DETAILED DESCRIPTION:
This was a phase 1, single-center study carried out in healthy male and female subjects to investigate the safety, tolerability, and PK of multiple doses (25mg, 50mg, and 75mg once daily) of d-methadone for 10 days. It was a double-blind, randomized, placebo-controlled study in sequential cohorts of healthy subjects. Subjects participated in the study for approximately 7 weeks. Eligible subjects were randomized within 30 days of screening. Of the 8 subjects in each cohort, 2 subjects received placebo and 6 subjects received d-methadone. The duration of dosing ensured that steady-state plasma concentrations were achieved.

A single ascending dose study previously conducted by Relmada Therapeutics, Inc. demonstrated that the maximum tolerated single dose for oral d-methadone in healthy opiate-naive subjects was 150 mg. The single doses of d-methadone appeared to be safe, with no indication of respiratory depression or clinically significant QTc prolongation, and minimal subjective pharmacodynamic (PD) effects.

The following assessments and procedures ensured the safety of the subjects during the study:

* continuous cardiac telemetry for 8 hours post-dose to detect any potential cardiac issues
* continuous pulse oximetry monitoring for 8 hours post-dose to detect any potential respiratory distress
* presence of a safety catheter to administer rescue medication (naloxone), if needed

The following signs of opioid toxicity were deemed to be of special interest:

* sustained respiratory depression that results in oxygen saturation below 92%
* QTc prolongation (>500 ms or >70 ms above the baseline)
* protracted nausea and vomiting
* any AE deemed by the investigator to be dose-limiting Safety Analysis Safety and tolerability parameters were listed by treatment and subject and displayed in summary tables using descriptive statistics. Original terms used to identify AEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 17.1. The number and percentage of subjects with treatment emergent AEs (TEAEs) were summarized by system organ class, preferred term, and treatment and for each treatment by maximum intensity and maximum relationship to study treatment.

Descriptive statistics for vital signs were calculated and presented for each time point by treatment group (absolute values and change from baseline). Safety ECG results were summarized using descriptive statistics; frequencies (numbers and percentages) were calculated for the overall evaluation by scheduled time and treatment group. Laboratory data were summarized by the type of test and scheduled visit. Descriptive statistics and number of subjects with laboratory test results below, within, and above normal ranges were tabulated by scheduled time. Abnormal findings in laboratory data were listed with a flag for clinical significance. Medical history abnormalities were coded to MedDRA terms and listed. Physical examination abnormalities were also listed. Data collected from the C-SSRS were classified into the Columbia Classification Algorithm of Suicide Assessment (C-CASA) categories and were listed. Frequency tables were used to summarize the total score from the COWS questionnaire, by treatment group. The original verbatim terms for concomitant medications were coded into drug class and preferred term. These data were listed.

Pharmacokinetic Analysis The PK parameters for d-methadone determined by non-compartmental analysis were summarized by dose. Graphs of concentration (linear and log-linear) vs time were generated. Descriptive statistics were calculated by dose and time point for all d-methadone concentrations. Concentrations below the limit of quantification (BLQ) were analyzed as outlined in the statistical analysis plan (SAP). Concentrations of l-methadone were analyzed only if the majority of values were not BLQ.

For the calculation of the PK parameters, concentration-time data were treated as follows: BLQ concentrations prior to the first quantifiable concentration were set to zero; BLQ concentrations after the first quantifiable concentration were treated as missing; pre-dose sampling times relative to dosing were set to zero. Descriptive statistics were calculated by dose. The dose proportionality of Cmax and AUC was assessed by the Hummel method. Tmax and t½ for different doses were compared using the Kruskal-Wallis test.

Pharmacodynamic Analysis The PD data at each time point were summarized by descriptive statistics and presented graphically (as appropriate). Derived endpoints were summarized using descriptive statistics. Pupillometry constriction was listed and grouped by treatment group and subject with descriptive statistics for changes from baseline for different time points.

Holter ECG Analysis (Cardiodynamic Analysis) The analysis of the Holter ECG data was performed using SAS®. The average of the 3 pre-dose time points on Day 1 was used as baseline for all post-dose time points. Heart rate and the PR, QRS, QT, and QTcF intervals collected from all randomized subjects were presented in data listings with the same precision as in the database. Data listings were sorted by treatment, subject number, day, and time point. Both absolute and change from baseline values for each subject were provided.

ELIGIBILITY:
Inclusion Criteria:

1. healthy male or female subjects, 18 to 55 years of age, inclusive
2. body mass index (BMI) within the range of 18.0 to 30.0 kg/m2, inclusive, and a minimum weight of 50.0 kg
3. non-smoker for at least 3 months and tested negative on a breath carbon monoxide (CO) test
4. male subjects of reproductive potential must have been using and willing to continue using medically acceptable contraception from screening and for at least 2 months after the last study drug administration
5. female subjects of childbearing potential must have been using and willing to continue using medically acceptable contraception for at least 1 month prior to screening (at least 3 months for oral, transdermal, vaginal ring contraceptives) and for at least 2 months after last study drug administration
6. female subjects of non-childbearing potential must have met the criteria defined in the clinical protocol
7. able to speak, read, and understand English sufficiently to allow completion of all study assessments
8. must have understood and provided written informed consent, prior to the initiation of any protocol-specific procedures

Exclusion Criteria:

1. self-reported substance or alcohol dependence (excluding nicotine and caffeine) within the past 2 years, and/or subjects who had ever been in a substance or alcohol rehabilitation program to treat their substance or alcohol dependence
2. subject-reported family history of substance abuse in an immediate family member (i.e., parent, sibling, or child)
3. history or presence of clinically significant abnormality as assessed by physical examination, medical history, 12-lead ECG, vital signs, or laboratory values, which in the opinion of the investigator would jeopardize the safety of the subject or the validity of the study results
4. chronic use of prescribed opioids (i.e., >120 days in a 6-month period) or any recreational use of opioids
5. evidence of clinically significant hepatic or renal impairment, including alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5× upper limit of normal (ULN) or bilirubin >1× ULN
6. history or family history of sudden unexplained death or long QT syndrome
7. QT interval corrected using Fridericia's formula (QTcF) >450 ms in females or >430 ms in males
8. history of hypotension
9. history or presence of any condition in which an opioid was contraindicated (e.g., significant respiratory depression, acute or severe bronchial asthma or hypercarbia, bronchitis, or had/was suspected of having paralytic ileus)
10. history of status asthmaticus, chronic pulmonary disease, or severe allergic reaction (including anaphylaxis) to any substance
11. use of an opioid within the 6 months prior to screening
12. use of a prohibited medication
13. positive urine drug screen
14. positive breath alcohol test; subjects with a positive result may have been rescheduled at the investigator's discretion
15. female subjects who were currently pregnant (had a positive pregnancy test)
16. history of allergy or hypersensitivity to methadone or related drugs (e.g., opioids)
17. positive for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
18. donation or loss of more than 500 mL of whole blood within 30 days prior to first drug administration
19. difficulty with venous access or unsuitable or unwilling to undergo catheter insertion
20. treatment with an investigational drug within 5 times the elimination half-life, if known (e.g., a marketed product) or within 30 days (if the elimination half-life is unknown) prior to first drug administration or was concurrently enrolled in any research judged not to be scientifically or medically compatible with this study
21. an employee of the sponsor or research site personnel directly affiliated with this study or their immediate family member, defined as a spouse, parent, sibling, or child, whether biological or legally adopted
22. a subject who, in the opinion of the investigator or designee, was considered unsuitable or unlikely to comply with the study protocol for any reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2015-11-16 (Actual); Study Completion 2015-11-16 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Change from pre-dose, Days 1 through 13, and Days 14, 16±1, and 18±1
  Spontaneously reported and observed AEs were recorded throughout the study, and AEs were elicited using a non-leading question at designated time points. Regardless of seriousness, intensity, or presumed relationship to study drug, all AEs were recorded in the source documentation from the time of first contact with the subject (e.g., screening) until the end of the follow-up period of the study. AEs that occurred after medical screening and prior to administration of the first dose of study drug were recorded in the source documentation as baseline signs and symptoms.

SECONDARY OUTCOMES:
Plasma levels | Days 1 through 13, and Days 14, 16±1, and 18±1
  Blood samples were collected to determine the plasma levels of d-methadone and l-methadone.

OTHER OUTCOMES:
Clinical Opiate Withdrawal Scale (COWS) | Days 11 through 13
  The Clinical Opiate Withdrawal Scale (COWS) is an 11-item scale designed to be administered by a clinician. This tool can be used in both inpatient and outpatient settings to reproducibly rate common signs and symptoms of opiate withdrawal and monitor these symptoms over time. The summed score for the complete scale can be used to help clinicians determine the stage or severity of opiate withdrawal and assess the level of physical dependence on opioids. The sum total of the 11 items are ranked by score. Score: 5- 1 2 = mild; 1 3-24 = moderate; 25-36 = moderately severe; more than 36 = severe withdrawal
Bond-Lader visual analog scale (VAS) assessment | Pre-dose and 3 hours post-dose on Day 1 to Day 10 and 72 hours post last dose
  The Bond-Lader visual analog scale (VAS) consists of 16 bipolar, self-rated, 101-point (from 0 to 100) scales between opposite adjectives. This VAS was adapted for computerized assessment. The subject had to indicate how they were feeling at the time of evaluation. Using a mouse, the subject positioned a cursor over a small vertical box (a "slider") and clicked on it to move it left or right on a horizontal line. To register the response, the subject had to press the "OK" button that appeared below the horizontal line.
Pupillometry | Pre-dose and 2, 4, 6, and 8 hours post-dose from Day 2 to Day 9, and from Day 10 to Day 13
  Pupillometry was used as an objective physiological PD measure as it is a sensitive measure of central opioid action and appears to be resistant to tolerance development with repeated administration. An electronic pupillometer was used to measure pupil diameter. Data from a series of frames were used in the calculation, and the final display showed the weighted average and standard deviation of the pupil size. Measurements were collected under mesopic lighting conditions.